CLINICAL TRIAL: NCT03392714
Title: Plasma and Cerebrospinal Fluid (CSF) Pharmacokinetics of Bendamustine as a Component of Salvage Therapy for Primary Central Nervous System Lymphoma (PCNSL)
Brief Title: Bendamustine-based Combination Therapy for PCNSL
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chonnam National University Hospital (Other)
Responsible Party: Principal Investigator, Deok-Hwan Yang, Principal Investigator, Chonnam National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CNUHH-2016-145
Record Dates: First submitted 2017-12-06; First posted 2018-01-08 (Actual); Last update posted 2018-01-08 (Actual); Status verified 2018-01

CONDITIONS: PCNSL
Keywords: Bendamustine; CSF; Pharmacokinetics; PCNSL; Salvage therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- R-B(O)AD (Experimental): Intravenous R-B(O)AD every 4 weeks for up to 4 cycles
  Interventions: Drug: R-B(O)AD

INTERVENTIONS:
Drug: R-B(O)AD — rituximab 375 mg/m2 on day 1; vincristine 1.4 mg/m2 on day 1, omitted in patients ≥70 years of age due to risk of neurotoxicity; bendamustine 75 mg/m2 over 1 h on days 2 and 3; cytarabine 1000 mg/m2 over 3 h on days 2-4; dexamethasone 20 mg on days 1-4, administered intravenously

SUMMARY:
This pilot study will i) evaluate the efficacy and the safety of bendamustine-based combination chemotherapy and ii) investigate the pharmacokinetics (PK)of bendamustine in plasma and CSF when given as salvage treatment for patients with relapsed or refractory primary central nervous system lymphoma (PCNSL).

DETAILED DESCRIPTION:
A relatively high proportion of patients diagnosed with primary CNS lymphoma will experience recurrent disease, yet therapy options are limited in salvage therapy. Based on the demonstrated activity and proposed additive mechanisms of the chemotherapeutic agents included in the bendamustine-based combination regimen, the efficacy and safety of R-B(O)AD will be evaluated for treatment of relapsed/refractory (R/R) primary CNS lymphoma. Evidence from previous preclinical tissue distribution studies and single agent intravenous drug therapy trials in CNS malignancies suggests that bendamustine penetrates brain and tumor tissue, however there are no clinical data available on the PK of bendamustine in the CSF. This study will evaluate the PK of plasma and CSF drug levels through a population based nonlinear mixed-effects model approach in a R/R PCNSL cohort with the goals to define the currently unknown PK profile of bendamustine in the CSF and to further characterize the relationship between plasma and CSF drug levels, and the influence of exposure on response to therapy.

ELIGIBILITY:
Inclusion Criteria:

1. PCNSL of diffuse large B-cell lymphoma (DLBCL) with a CNS lesion by tissue biopsy
2. Age ≥ 19 years old
3. Relapsed or refractory PCNSL after frontline combined chemotherapy or radiation
4. ECOG performance status 0-2
5. Absolute neutrophil count ≥ 1000/uL
6. Platelets ≥ 100,000/uL
7. Total bilirubin ≤ 1.5 x ULN (upper limit of normal)
8. Aspartate aminotransferase (AST) ≤ 3 x ULN
9. Creatinine ≤ 2.0 x ULN

Exclusion Criteria:

1. PCNSL of other than DLBCL or T-cell lymphoma with a CNS lesion by tissue biopsy
2. Any of the following: pregnant women, nursing women, men or women of childbearing potential who are unwilling to employ adequate contraception
3. Uncontrolled infection
4. Therapy with myelosuppressive chemotherapy or biologic therapy < 21 days prior to registration
5. Persistent toxicities ≥ grade 3 from prior chemotherapy or biologic therapy regardless of interval since last treatment
6. History of thromboembolic episodes ≤ 3 months prior to registration
7. Active hepatitis B or C with uncontrolled disease
8. Active other malignancy requiring treatment that would interfere with the assessments of response of the lymphoma to protocol treatment
9. Any severe and/or uncontrolled medical conditions or other conditions that could adversely impact their ability to participate in the study
10. Major surgery ≤ 4 weeks prior to registration or have not recovered from side effects of such therapy

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2016-01-20 (Actual); Primary Completion 2018-01-20 (Estimated); Study Completion 2019-01-20 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | 2 year
  rate of complete or partial response (CR/PR)

SECONDARY OUTCOMES:
Toxicity based on NCI Common Terminology Criteria version 4.0 | 2 year
  adverse event incidence of combination regimen
Progression-free survival (PFS) | 2 years
  calculated from the time of study entry until progression, relapse, or death
Overall survival (OS) | 2 years
  calculated from the time of study entry until death
Maximum concentration [Cmax] of bendamustine in plasma and CSF | 6 months
  peak concentration of bendamustine after 1 hour IV infusion
Area under the curve [AUC] of bendamustine in plasma and CSF | 6 months
  overall exposure of bendamustine after IV infusion

CONTACTS AND LOCATIONS:
Overall Officials: Deok-Hwan Yang, MD, Principal Investigator — Chonnam National University Hwasun Hospital, Department of Hematology-Oncology
Locations (1):
- Chonnam National University Hwasun Hospital, Hwasun-gun, Jeollanam-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim T, Choi HY, Lee HS, Jung SH, Ahn JS, Kim HJ, Lee JJ, Yoo HD, Yang DH. Clinical response and pharmacokinetics of bendamustine as a component of salvage R-B(O)AD therapy for the treatment of primary central nervous system lymphoma (PCNSL). BMC Cancer. 2018 Jul 9;18(1):729. doi: 10.1186/s12885-018-4632-y. PMID 29986691